CLINICAL TRIAL: NCT02239354
Title: A Prospective, Multicenter, Open-Label, First-in-Human Phase 1/2 Study With Two Cohorts to Evaluate the Safety, Tolerability, and Efficacy of Various Doses of VC-01™ Combination Product in Subjects With Type 1 Diabetes Mellitus
Brief Title: A Safety, Tolerability, and Efficacy Study of VC-01™ Combination Product in Subjects With Type I Diabetes Mellitus
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Insufficient functional product engraftment
Sponsor: ViaCyte (Industry)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: VC01-101
Record Dates: First submitted 2014-09-09; First posted 2014-09-12 (Estimated); Results first posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-02

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

ARMS (2):
- Cohort 1 (Experimental): 2 VC-01™ Combination Product implants
  Interventions: Combination Product: VC-01™ Combination Product
- Cohort 2 (Experimental): 4 or 6 VC-01™ Combination Product implants
  Interventions: Combination Product: VC-01™ Combination Product

INTERVENTIONS:
Combination Product: VC-01™ Combination Product — Biologic and Device

SUMMARY:
The purpose of this trial is to test if VC-01™ combination product can be implanted subcutaneously in subjects with Type 1 Diabetes and maintained safely for two years. It will also test if VC-01 is an effective treatment for subjects with Type 1 Diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Men and women (non-pregnant and non-childbearing potential)
* Diagnosis of type 1 diabetes mellitus for at least 3 years
* Stable diabetic treatment
* Willingness to use a continuous glucose meter
* Acceptable candidate for implantation

Exclusion Criteria:

* Advanced complications associated with diabetes
* Immunosuppressive therapy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- University of California at San Diego, San Diego, California, United States
- University of Alberta Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Satin LS, Soleimanpour SA, Walker EM. New Aspects of Diabetes Research and Therapeutic Development. Pharmacol Rev. 2021 Jul;73(3):1001-1015. doi: 10.1124/pharmrev.120.000160. PMID 34193595
- [Derived] Saber N, Bruin JE, O'Dwyer S, Schuster H, Rezania A, Kieffer TJ. Sex Differences in Maturation of Human Embryonic Stem Cell-Derived beta Cells in Mice. Endocrinology. 2018 Apr 1;159(4):1827-1841. doi: 10.1210/en.2018-00048. PMID 29420708
- [Derived] Pase C, Mathias AD, Garcia CD, Garcia Rodrigues C. Using Social Media for the Promotion of Education and Consultation in Adolescents Who Have Undergone Kidney Transplant: Protocol for a Randomized Control Trial. JMIR Res Protoc. 2018 Jan 9;7(1):e3. doi: 10.2196/resprot.8065. PMID 29317381

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Up to 2 VC-01-250™ Combination Product implants
  Up to 6 VC-01-20 sentinel units
  VC-01™ Combination Product: Biologic and Device
- Cohort 2: Up to 4 or 6 VC-01™ Combination Product implants
  Up to 3 VC-01-20 sentinel units
  VC-01™ Combination Product: Biologic and Device
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 19 | 0
Completed | 9 | 0
Not Completed | 10 | 0

BASELINE CHARACTERISTICS:
Population: Cohort 2 enrollment was never initiated and is therefore 'zero'.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 19 | 0 | 19
Age, Continuous [Median (Standard Deviation); unit: years] | 29.0 (11.92) |  | 29.0 (11.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 18 |  | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 |  | 1
  Not Hispanic or Latino | 18 |  | 18
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 19 |  | 19
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events Reported During the Study.
Time Frame: Thru the Month 24 Visit
Population: The Safety Analysis Set (SAS) will include all T1DM subjects who were enrolled into the study and in whom an implant surgery was attempted, regardless if any VC-01-250 units or sentinel-sized units were actually implanted. This includes all subjects in both Cohort 1 and Cohort 2.
Measure: Number; unit: events
Arm/Group | Cohort 1
Number analyzed (Participants) | 19
events | 114

2. Primary Outcome: Change in C-peptide
Description: The Full Analysis Set (FAS) is the intent-to-treat (ITT) set of subjects. This set is defined as all T1DM subjects who were enrolled into the study and received implantation of at least one VC-01-250 or sentinel unit on Study Day 1. The FAS (Cohort 2 T1DM subjects who meet the FAS criteria) will be used to analyze the primary efficacy endpoint.
Time Frame: Baseline to the Month 6 Visit
Population: No subjects were enrolled in Cohort 2. Therefore, no data was collected for this endpoint.
Arm/Group | Cohort 2
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: AEs are recorded on the CRF from Visit 2 (Week-3) through the last subject visit (out to two years). At the conclusion of the trial, any ongoing AEs were followed up for 28 days after the explantation procedure.
Description: All observed or volunteered AEs regardless of suspected causal relationship to the investigational product were reported. For all AEs, the Investigator obtained information adequate to determine the outcome of the AE, whether it meets the criteria for classification as a serious adverse event(SAE), the causality, and the severity,
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/0
Serious Adverse Events (participants affected / at risk) | 2/19 | 0/0
Other Adverse Events (participants affected / at risk) | 18/19 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=19) | Cohort 2 (N=0)
Cellulitis (Infections and infestations) | 1 (1) | NA
Right middle lobe pneumonia (Infections and infestations) | 1 (1) | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=19) | Cohort 2 (N=0)
Procedural pain (Injury, poisoning and procedural complications) | 14 (30) | NA
Contusion (Injury, poisoning and procedural complications) | 2 (2) | NA
Incision site haematoma (Injury, poisoning and procedural complications) | 2 (2) | NA
Post procedural haematoma (Injury, poisoning and procedural complications) | 2 (2) | NA
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | NA
Post procedural inflammation (Injury, poisoning and procedural complications) | 1 (1) | NA
Post procedural swelling (Injury, poisoning and procedural complications) | 1 (1) | NA
Procedural complication (Injury, poisoning and procedural complications) | 1 (1) | NA
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | NA
Venous injury (Injury, poisoning and procedural complications) | 1 (1) | NA
Wound (Injury, poisoning and procedural complications) | 1 (1) | NA
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | NA
Device dislocation (General disorders) | 7 (10) | NA
Device breakage (General disorders) | 5 (5) | NA
Implant site extravasation (General disorders) | 5 (7) | NA
Implant site haemorrhage (General disorders) | 2 (3) | NA
Implant site hypoaesthesia (General disorders) | 2 (2) | NA
Implant site swelling (General disorders) | 2 (2) | NA
Calcinosis (General disorders) | 1 (1) | NA
Complication of device removal (General disorders) | 1 (1) | NA
Device difficult to use (General disorders) | 1 (1) | NA
Device extrusion (General disorders) | 1 (1) | NA
Implant site oedema (General disorders) | 1 (1) | NA
Implant site pain (General disorders) | 1 | NA
Implant site rash (General disorders) | 1 (1) | NA
Localised oedema (General disorders) | 1 (1) | NA
Oedema peripheral (General disorders) | 1 (1) | NA
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (2) | NA
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | NA
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | NA
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | NA
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | NA
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | NA
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | NA
Anaemia (Blood and lymphatic system disorders) | 1 (1) | NA
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | NA
White blood cell disorder (Blood and lymphatic system disorders) | 1 (1) | NA
Nausea (Gastrointestinal disorders) | 3 (3) | NA
Constipation (Gastrointestinal disorders) | 2 (2) | NA
Vomiting (Gastrointestinal disorders) | 2 (2) | NA
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | NA
Diarrhoea (Gastrointestinal disorders) | 1 (1) | NA
Cellulitis (Infections and infestations) | 2 (2) | NA
Pneumonia (Infections and infestations) | 1 (1) | NA
Wound infection (Infections and infestations) | 1 (1) | NA
Hypoaesthesia (Nervous system disorders) | 1 (1) | NA
Paraesthesia (Nervous system disorders) | 1 (1) | NA
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA
Sensitisation (Immune system disorders) | 1 (1) | NA
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | NA
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | NA

LIMITATIONS AND CAVEATS:
Study did not proceed to Cohort 2 to evaluate efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multi-center publication is not published within 14 to 18 months (depends on the individual PI's contract) after completion of the study, the PI will have the right to publish and present results. The PI will submit any proposed publication or presentation to the Sponsor for review at least 30 to 60 days (depending on the individual PI's contract) prior to submitting any such proposed publication to a publisher, proceeding with such proposed presentation or making any other disclosure.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-01): https://cdn.clinicaltrials.gov/large-docs/54/NCT02239354/Prot_SAP_000.pdf